CLINICAL TRIAL: NCT00156676
Title: Pilot Study on Gait & Motor Function in MS Using BWS Treadmill Training
Brief Title: Restoration of Walking in Multiple Sclerosis Using Treadmill Training.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B4031-I; NCT00127426 (obsolete NCT alias)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Multiple Sclerosis
Keywords: Disability; Gait; Multiple Sclerosis; Rehabilitation; Robot
MeSH Terms: conditions — Multiple Sclerosis

ARMS (2):
- Arm 1 (Experimental): Cross over from body-weight support treadmill to Lokomat
  Interventions: Device: Body-weight supported treadmill; Device: Lokomat
- Arm 2 (Experimental): Cross over from Lokomat to body-weight support treadmill
  Interventions: Device: Body-weight supported treadmill; Device: Lokomat

INTERVENTIONS:
Device: Body-weight supported treadmill
  Arms: Arm 1
Device: Lokomat
  Arms: Arm 1
Device: Body-weight supported treadmill
  Arms: Arm 2
Device: Lokomat
  Arms: Arm 2

SUMMARY:
The primary purpose of this study is to collect preliminary and pilot data to begin to determine whether the use of body weight support treadmill therapy (BWSTT) with and without driven-gait-orthotics (DGO), results in improved motor recovery and ambulation MS patients with gait impairment

DETAILED DESCRIPTION:
Gait impairment is a major cause of ongoing disability in patients with multiple sclerosis (MS). New treadmills that provide body weight support and even robotic assistance to the lower limbs have recently been developed and are now commercially available. These treadmills allow the subject to execute the integrated process of walking in a task-specific manner that is repetitively reinforced in a normal pattern. Data from studies using these body-weight supported treadmills (BWSTT) in spinal cord injury and stroke patients suggest that intensive task-specific gait rehabilitative training may help to restore a normative gait pattern, improve overground walking and enhance quality of life in multiple sclerosis patients with neurological gait impairment. In this study, we propose a series of prospective longitudinal clinical studies to collect pilot data on the use of task-specific BWSTT +/- Lokomat on improving ambulation, motor function and quality of life for MS patients with mild to moderate gait difficulty. Pilot data will also be collected for the effect conventional rehabilitation has on ambulation and motor outcomes as well as how these outcomes change during usual care. Our clinical research goals are to capture the initial pilot data (mean changes and variances in ambulation, motor, fatigue and quality of life outcomes) to facilitate the design of a larger clinical trial to test efficacy if these preliminary data are promising. The planned studies will study the effect of two forms of task specific training (BWSTT alone and BWSTT combined with Lokomat) compared to conventional gait rehabilitative methods and usual care

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MS by McDonald criteria. EDSS level between 4-6.5.

Exclusion Criteria:

* Cardiovascular: recent MI < 4 wk, uncontrolled HTN >190/110 mmHg, Uncontrolled diabetes (blood glucose 2X above the upper limit of normal or non-fasting blood drain).
* Symptomatic fall in blood pressure (>30mm Hg), when upright in the body support apparatus, despite medical therapy.
* Circulatory problems, history of vascular claudication or pitting edema.
* Cognitive impairment MMSE < 21.
* Body weight over 150 kg (structural limits of the Lokomat).
* Lower extremity injuries that limit range of motion or function.
* Joint problems (hip or leg) that limit range of motion or cause pain with movement despite treatment.
* Unstable fractures.
* Pressure sores with any skin breakdown in areas in contact with the body harness or DGO apparatus.
* Chronic and ongoing alcohol or drug abuse.
* Pre-morbid, ongoing depression or psychosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Mean changes and variances in ambulation, motor, fatigue and quality of life | Baseline, cross-over, study endpoint
  Timed 25 foot walk

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lo, MD PhD, Principal Investigator — Providence VA Medical Center
Locations (1):
- Providence VA Medical Center, Providence, Rhode Island, United States

REFERENCES:
- [Result] Lo AC, Triche EW. Improving gait in multiple sclerosis using robot-assisted, body weight supported treadmill training. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):661-71. doi: 10.1177/1545968308318473. PMID 18971381
- [Derived] Wier LM, Hatcher MS, Triche EW, Lo AC. Effect of robot-assisted versus conventional body-weight-supported treadmill training on quality of life for people with multiple sclerosis. J Rehabil Res Dev. 2011;48(4):483-92. doi: 10.1682/jrrd.2010.03.0035. PMID 21674396